CLINICAL TRIAL: NCT07372950
Title: Randomized Controlled Trial of Different Behavioral Text Messages to Improve Influenza Vaccination Rates
Brief Title: Kaiser Colorado Flu Nudge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Michael Ho, Medical Director of IMPROVE, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2368690-1
Record Dates: First submitted 2025-10-01; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Influenza; Vaccination
Keywords: influenza; vaccination; text messages; behavioral change
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Generic text messages (Active Comparator): Patients will receive the usual flu vaccine text message reminder
  Interventions: Behavioral: Behavioral economics framed test messaging
- Positively framed (Experimental): Patients will receive a positively framed text message to get the flu vaccine
  Interventions: Behavioral: Behavioral economics framed test messaging
- Convenience framed (Experimental): Patients will receive a convenience framed text message to get the flu vaccine
  Interventions: Behavioral: Behavioral economics framed test messaging

INTERVENTIONS:
Behavioral: Behavioral economics framed test messaging — We will use positive framing and convenience framing as our 2 behavioral text messages to improve flu vaccination rates.

SUMMARY:
Influenza infection leads to significant morbidity and mortality each year. Influenza vaccines can reduce the risk of flu and the severity of flu illness, In addition, flu vaccinations can reduce flu complications such as pneumonia or worsening of chronic heart or lung disease. Each year, Kaiser Permanente of Colorado offers influenza vaccines to patients at no cost either at primary care clinic appointments or flu walk-in clinics in the fall prior to the upcoming flu season. In addition, as part of clinic appointment reminder text messages, there is a message to get the flu vaccine for patients who have not received the vaccine prior to the clinic visit. Building on these flu reminder text messages for patients who have not received a flu vaccine, this study will test different behavioral nudge text messages to improve influenza vaccination rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients 6 months and older who have not received a flu shot at the time of their primary care clinic appointment reminder will be eligible to receive a flu vaccine reminder text message. For children <18 years of age, their caregiver will receive the text message

Exclusion Criteria:

* Patients not eligible for flu vaccine

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Receive flu vaccine | 12 weeks following receipt of first text message reminder
  Did the patient receive a flu vaccine as denoted from the EMR. The vaccine could have occurred within Kaiser Permanente Colorado or outside of Kaiser Permanente Colorado and in which Kaiser received information about the flu vaccination during the flu season 2025-2026.

SECONDARY OUTCOMES:
Time to flu vaccination | 12 weeks following receipt of 1st text message reminder
  Time from primary care clinic visit that triggered the flu reminder text message and date of flu vaccination as denoted in the EMR.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ho, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Institute for Health Research, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No